CLINICAL TRIAL: NCT00016263
Title: Randomized Study Of Dacarbazine Versus Dacarbazine Plus G3139 (Bcl-2 Antisense Oligonucleotide) In Patients With Advanced Malignant Melanoma
Brief Title: Dacarbazine With or Without Oblimersen (G3139) in Treating Patients With Advanced Malignant Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genta Incorporated (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068616; GENTA-GM301; UCLA-0207109
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2002-10

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — oblimersen; Dacarbazine

INTERVENTIONS:
Biological: oblimersen sodium
Drug: dacarbazine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Oblimersen (G3139) may help dacarbazine kill more cancer cells by making tumor cells more sensitive to the drug. It is not yet known if dacarbazine is more effective with or without oblimersen (G3139).

PURPOSE: Randomized phase III trial to compare the effectiveness of dacarbazine with or without oblimersen (G3139) in treating patients who have advanced malignant melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the survival of patients with advanced malignant melanoma treated with dacarbazine with or without oblimersen (G3139).
* Compare the response rate, durable response rate, and progression-free survival of patients treated with these regimens.
* Compare the safety of these regimens in this patient population.
* Compare the performance status, body weight, and tumor-related symptoms of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to ECOG performance status (0 vs 1 or 2), extent of metastases and lactate dehydrogenase (LDH) level (skin subcutaneous and/or lymph node metastases without visceral involvement and normal LDH vs any visceral metastases or elevated LDH), and liver metastases (yes vs no). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive dacarbazine IV over 60 minutes on day 1.
* Arm II: Patients receive oblimersen (G3139) IV continuously over days 1-6 followed by dacarbazine IV over 60 minutes on day 6.

Treatment repeats every 21 days for a maximum of 8 courses in the absence of disease progression or unacceptable toxicity. Patients with stable disease or partial or complete response may be eligible for another 8 courses of treatment in an extension protocol.

Patients are followed at least every 2 months for up to 2 years after study.

PROJECTED ACCRUAL: A total of 750 patients (375 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant melanoma

  * Progressive disease that is unresectable or metastatic
* No primary ocular or mucosal melanoma
* At least 1 unidimensionally measurable lesion by physical exam or imaging studies

  * At least 10 mm by caliper for superficial cutaneous disease
  * At least 20 mm by contrast-enhanced or spiral CT scan for visceral or nodal/soft tissue disease
  * No bone metastases as only site of measurable disease
  * Lesions considered non-measurable include the following:

    * Bone lesions
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging
    * Lesions located in a previously irradiated area
* No brain metastases or leptomeningeal disease
* Considered a medical candidate for dacarbazine treatment

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8 g/dL (hematopoietic growth factor or transfusion independent)

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT/AST no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* Albumin at least 2.5 g/dL
* PT/PTT no greater than 1.5 times ULN
* No history of chronic hepatitis or cirrhosis

Renal:

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* No uncontrolled congestive heart failure
* No New York Heart Association class III or IV disease
* No symptomatic coronary artery disease (e.g., uncontrolled arrhythmias or recurrent chest pain despite prophylactic medication)
* No cardiovascular signs and symptoms at least grade 2 within the past 4 weeks

Other:

* Intellectually, emotionally, and physically able to maintain an ambulatory infusion pump
* Satisfactory venous access
* No other significant medical disease
* No uncontrolled seizure disorder
* No active infection
* No uncontrolled diabetes mellitus
* No active autoimmune disease
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No known hypersensitivity to phosphorothioate-containing oligonucleotides or dacarbazine
* No known HIV infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy, cytokine, biologic, or vaccine therapy in the adjuvant and/or metastatic setting and recovered
* No concurrent prophylactic growth factors (e.g., filgrastim [G-CSF], sargramostim [GM-CSF] or epoetin alfa) during course 1 of study

Chemotherapy:

* No prior cytotoxic chemotherapy, including regional perfusion

Endocrine therapy:

* No concurrent chronic corticosteroids with an average dose of at least 20 mg of prednisone or equivalent per day

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy to measurable target lesions unless progression occurred at that site or measurable disease developed outside the treated area

Surgery:

* At least 4 weeks since prior surgery and recovered
* No prior organ allografts

Other:

* At least 3 weeks since prior experimental therapy
* No prior intratumoral injection therapy to measurable target lesions unless progression occurred at that site or measurable disease developed outside the treated area
* No concurrent immunosuppressive drugs
* No concurrent anticoagulation therapy except 1 mg/day of warfarin for central line prophylaxis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-07; Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley R. Frankel, MD, Study Chair — Genta Incorporated
Locations (2):
- United States (2):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Genta Incorporated, Berkeley Heights, New Jersey